CLINICAL TRIAL: NCT00218998
Title: Effective Endurance Training in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Training in metabolic syndrome
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Impaired Glucose Tolerance; Overweight; Hypertension; Dyslipidemia
Keywords: Exercise; Exercise therapy
MeSH Terms: conditions — Glucose Intolerance; Overweight; Hypertension; Dyslipidemias; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: exercise training

SUMMARY:
To see how fast and how much physical training can reduce risk factors related to metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* insulin resistance, impaired glucose tolerance or type 2-diabetes, including two or more of the following factors: Blood pressure ≥ 140/90 mm Hg, Triglycerides Fasting ≥ 1,7 mmol/l, and/or low HDL-cholesterol (≤ 0,9 mmol/l in men, ≤ 1,0 mmol/l in women)
* Obesity, Waist-hip ratio ≥ 0,9 in men, ≥ 0,85 in women or BMI (body mass index) ≥ 30 kg/m2
* Microalbuminuria (albumin secretion ≥ 20 mg/l or 20 - 200 g per minute)

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-01 (Actual)

PRIMARY OUTCOMES:
To reduce risk factors related to metabolic syndrome

SECONDARY OUTCOMES:
Improve endothelial functions in patient with metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik E Wisløff, Phd prof, Study Chair — National Taiwan Normal University
Locations (1):
- The medical faculty at norwegian university of science and technology, Trondheim, Norway

REFERENCES:
- [Background] Poelkens F, Hopman MT, Tack CC. Letter by Poelkens et al regarding article, "Aerobic interval training versus continuous moderate exercise as a treatment for the metabolic syndrome: a pilot study". Circulation. 2009 Mar 3;119(8):e225; author reply e226. doi: 10.1161/CIRCULATIONAHA.108.818765. No abstract available. PMID 19255350
- [Result] Tjonna AE, Lee SJ, Rognmo O, Stolen TO, Bye A, Haram PM, Loennechen JP, Al-Share QY, Skogvoll E, Slordahl SA, Kemi OJ, Najjar SM, Wisloff U. Aerobic interval training versus continuous moderate exercise as a treatment for the metabolic syndrome: a pilot study. Circulation. 2008 Jul 22;118(4):346-54. doi: 10.1161/CIRCULATIONAHA.108.772822. Epub 2008 Jul 7. PMID 18606913